CLINICAL TRIAL: NCT06138886
Title: Calisthenics Exercise Program and Pulsed Electromagnetic Therapy on Liver Function Following Burn Injuries.
Brief Title: Calisthenics Exercise and Electromagnetic Therapy on Liver Function Following Burn Injuries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Gamal Fawzy El-Sayed, Lecturer of physical therapy of surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004650
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Burns
Keywords: Elevated plasma liver enzymes
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Calisthenics exercise group (Experimental): This group includes 30 burned patients who will perform calisthenics exercises program for 3 months (3 times/week) in addition to their traditional physical therapy program and medical treatment.
  Interventions: Other: calisthenics exercises
- Pulsed electromagnetic therapy group (Experimental): This group includes 30 burned patients who will receive pulsed electromagnetic therapy for 3 months (3 times/week) in addition to their traditional physical therapy program and medical treatment.
  Interventions: Device: Pulsed electromagnetic therapy
- Calisthenics exercises and pulsed electromagnetic therapy group (Experimental): This group includes 30 burned patients who will perform calisthenics exercises program and receive pulsed electromagnetic therapy for 3 months (3 times/week) in addition to their traditional physical therapy program and medical treatment.
  Interventions: Device: Pulsed electromagnetic therapy; Other: calisthenics exercises

INTERVENTIONS:
Device: Pulsed electromagnetic therapy — The appliance will be connected to electrical mains supplying 230V± 10%. The solenoids are adjusted to be over the upper abdominal area. The options of the appliance are adjusted with very low frequency (15 HZ), very low intensity (20 G) for 20 minutes, and 3 sessions / week for successive 3 months.
  Arms: Calisthenics exercises and pulsed electromagnetic therapy group; Pulsed electromagnetic therapy group
Other: calisthenics exercises — This group includes 30 burned patients who will perform calisthenics exercises program for 3 months (3times/week) in addition to their traditional physical therapy program and medical treatment.
  Arms: Calisthenics exercise group; Calisthenics exercises and pulsed electromagnetic therapy group

SUMMARY:
Serum concentrations of alanine transaminase (ALT) and aspartate transaminase (AST) significantly increased immediately upon burn trauma and remained significantly elevated for about three years.

Calisthenics exercises consist of movements that increase the flexibility and strength of the body. It is a type of exercise consisting of various movements applied without equipment and apparatus, using your body weight.

Clinical evidence shows that PEMF therapy reduces pain associated with trauma from accidents, sports injuries, surgeries and burns as well as from disease and degeneration. PEMF therapy improves these conditions in many different concurrent ways including mechanical, chemical, electrical and magnetic processes within the cells of the body.

DETAILED DESCRIPTION:
-Measurement procedures: Serum blood draws will be taken by certified technicians with the participant in a seated position.

Spectrophotometry is the measurable analysis technique using electromagnetic spectra. It deals with the ranges of wavelengths such as near ultraviolet, near-infrared and visible light. A device called a spectrophotometer is used to measure the absorbance or transmittance through a liquid sample. The spectrophotometer measures a specific wavelength and it is possible to choose any wavelength in the spectrophotometer register as the double beam sends a beam through a blank reference sample and one through the sample to be measured.

Normal values that will be used for patients are 0-45 IU/l for Alanine transaminase (ALT) and 0-35 IU/l for Aspartate transaminase(AST).

Measurements will be taken before the treatment (pre-treatment) and after 3 months (post-treatment).

2-Therapeutic procedures: 2. a: Procedures of calisthenics exercises program: The workout schedule will last for 12 weeks with medium-intensity calisthenics exercises of 60 minutes for 3 days in a week. The intensity will be held at the pace at which the participants feel comfortable. In each workout period, after 10 minutes of warm-up, the exercises will be done in 45 minutes as pistol squat, leg raise, lunge stop, Russian twist, shoulder taps, inverse pull-up, dips, supermen exercise and crunch for 3 sets/8 repetitions and plank exercise for 3 sets/30min. Every workout will end with 5 minutes of cooling exercises.

2. b: Procedures of Pulsed electromagnetic therapy: The treatment procedures will start after the patient's release from the intensive care unit.

The patient will be asked to remove metal objects or anything sensitive to the magnetic field such as chains, belts, watches, etc.… before lying on the bed. Then the patient will be in a comfortable supine lying position over the motorized bed. During application, the patient will be asked not to move and remain stable as much as possible. The appliance will be connected to electrical mains supplying 230V± 10%. The solenoids are adjusted to be over the upper abdominal area. The options of the appliance are adjusted with very low frequency (15 HZ), very low intensity (20 G) for 20 minutes, 3 sessions/week for successive 3 months

ELIGIBILITY:
Inclusion Criteria:

* Age ranges between 20-45 years.
* Male and female patients will participate in the study.
* All patients have burns with BBSA about 30% to 50%
* All patients enrolled on the study will have their informed consent

Exclusion Criteria:

* Cardiac diseases.
* Burn of the sole of foot.
* Exposed hand or foot tendons.
* Upper or Lower limb amputation.
* History of liver diseases.
* Body mass index (BMI=kg/cm2)<30%.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Concentration of Alanine transaminase (ALT) and Aspartate transaminase(AST) enzymes in blood plasma. | Three months
  Liver enzymes

CONTACTS AND LOCATIONS:
Overall Officials: A G Elsayed, PHD, Study Chair — Cairo University
Locations (1):
- Faculty of Physical therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No